CLINICAL TRIAL: NCT04428346
Title: A Pilot Two-arm, Individual-level, Randomised Controlled Trial to Assess the Effect of an Intervention Integrating Contingency Management (Financial Incentives) to Enhance Hepatitis C Treatment Uptake Following Dried Blood Spot Hepatitis C RNA Testing Among People With Recent Injecting Drug Use Attending Needle and Syringe Programs
Brief Title: A Trial to Assess the Effect of an Intervention Integrating Contingency Management (Financial Incentives) to Enhance Hepatitis C Treatment Uptake Following Dried Blood Spot Hepatitis C RNA Testing Among People With Recent Injecting Drug Use Attending Needle and Syringe Programs
Acronym: AMPLIFY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: VHCRP2004
Record Dates: First submitted 2020-05-10; First posted 2020-06-11 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Participants will be randomised with a computerised random number generator (or random number table) with block randomisation to assist with keeping participant balance between study arms with a small sample size.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contigency Management (Intervention) (Active Comparator)
  Interventions: Behavioral: Incentive payment
- Standard of Care (Control) (No Intervention)

INTERVENTIONS:
Behavioral: Incentive payment — Incentive payment to enhance HCV treatment uptake among people with recent injecting drug use attending needle and syringe programs.
  Arms: Contigency Management (Intervention)

SUMMARY:
A pilot two-arm, individual-level, randomised controlled trial to assess the effect of an intervention integrating contingency management (financial incentives) to enhance hepatitis C treatment uptake following dried blood spot hepatitis C RNA testing among people with recent injecting drug use attending needle and syringe programs: the AMPLIFY study

ELIGIBILITY:
Inclusion Criteria:

1. Participants have voluntarily signed the informed consent form
2. 18 years of age or older
3. Recent injecting drug use (previous six months)

Exclusion Criteria:

1) Inability or unwillingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants who initiate Hepatitis C Virus treatment within 12 weeks of testing | 6 months
  Data will be presented in percentages and mean (SD) or median values (interquartile range), as appropriate. Chi square test or Fisher's exact test will be utilised, as appropriate, to examine between group differences.

SECONDARY OUTCOMES:
Feasibility of recruitment through a peer-based referral incentivization scheme | 6 months
  Recruitment numbers
Time to HCV treatment initiation | 6 months
Time to HCV treatment completion | 6 months
Time to visit to confirm viral cure (e.g. sustained virological response, SVR12) | 6 months
Participant perceptions and acceptability of being involved in a contingency management study will be assessed by study questionnaire | 6 months
Feasibility of a contingency management intervention to enhance hepatitis C treatment uptake | 6 months
  Proportion of participants who enrolled in the study and where assigned treatment who commenced treatment.

IPD SHARING:
Plan to Share IPD: No